CLINICAL TRIAL: NCT06528184
Title: Evaluating the Impact of Different Methods of HPV DNA Testing for Cervical Cancer Screening in Primary Care Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: National Healthcare Group, Singapore (Other Government); KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Ng Xin Rong, Family Physician, National Healthcare Group Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/00194; SCS-GRA-2023-00253 (Other Grant/Funding Number: Singapore Cancer Society)
Record Dates: First submitted 2024-07-03; First posted 2024-07-30 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care arm (Active Comparator): Participants will only be offered clinician-sampling for HPV DNA testing to determine if they are agreeable to undergo screening.
  Interventions: Diagnostic Test: Clinician-sampled HPV DNA test
- Intervention arm (Experimental): Participants will be offered clinician-sampling or self-sampling for HPV DNA testing to determine if they are agreeable to undergo screening using either modality.
  Interventions: Diagnostic Test: Self-sampled HPV DNA testing; Diagnostic Test: Clinician-sampled HPV DNA test

INTERVENTIONS:
Diagnostic Test: Self-sampled HPV DNA testing — Participants will be offered HPV DNA testing done through self-sampling (using self-sampling HPV DNA kits to obtain a mid-vaginal swab)
  Arms: Intervention arm
Diagnostic Test: Clinician-sampled HPV DNA test — Participants will be offered HPV DNA testing through clinician sampling (clinician-sampling (speculum examination by a nurse to obtain a cervical swab)

SUMMARY:
Primary objective of the study is to determine the extent that offering of self-sampling in addition to clinician-sampling Human Papillomavirus (HPV) DNA testing will increase detection of HPV DNA through an increase in uptake rates of cervical cancer screening as compared to offering clinician-sampling HPV DNA testing alone.

The hypothesis is that offering additional self-sampling will increase the detection of high-risk HPV DNA by at least 7.7%.

DETAILED DESCRIPTION:
This study is a pragmatic, multi-center, 1:1 randomized controlled trial designed to evaluate the impact of self-sampling HPV DNA testing on clinical outcomes and cost-effectiveness in cervical cancer screening. The trial will compare 2 approaches to HPV DNA testing within public primary care settings.

Participants in the intervention arm will first be offered a clinician-sampling HPV DNA test. If they decline, they will be offered the option of self-sampling HPV DNA test. The control arm will follow the standard protocol of offering only the conventional clinician-sampling HPV DNA test, reflecting the current standard of care in cervical cancer screening.

This study seeks to provide robust evidence on whether self-sampling can improve clinical outcomes, be cost-effective and be feasibility implemented in routine public primary healthcare settings. The findings are expected to inform future guidelines and policies for cervical cancer screening programs.

ELIGIBILITY:
Inclusion Criteria:

* 30-69 years old female Singapore citizens
* Due for cervical cancer screening
* Engaged in sexual intercourse before
* Able to give informed consent
* Able to read and communicate in English, Chinese or Malay

Exclusion Criteria:

* Virgo intacta
* Pregnancy
* History of cervical cancer, precancerous cervical lesions and total hysterectomy

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 650 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of high-risk Human Papillomavirus (HPV) DNA | 3 months
  Difference in detection of high-risk HPV DNA between 2 arms

SECONDARY OUTCOMES:
Uptake of cervical cancer screening | 3 months
  Difference in uptake of cervical cancer screening between 2 arms. Based on the number of cervical cancer screening tests that are processed and have available results.
Colposcopy referrals | 2 years
  Difference in colposcopy referrals between 2 arms. Based on the number of colposcopy referrals made to the tertiary hospital for abnormal cervical cancer screening test results in either arm.
Detection of cervical intraepithelial neoplasia (CIN) 2, CIN 3 and cervical cancers | 2 years
  Difference in detection of CIN 2, CIN 3 and cervical cancers between both arms.
Treatments for CIN 2, CIN 3 and cervical cancers | 2 years
  Difference in treated CIN 2, CIN 3 and cervical cancers between both arms. Based on the number of participants with CIN 2, CIN 3 and cervical cancers that have undergone treatments by a gynecologist in either arm.
Cost-effectiveness of cervical cancer screening | 2 years
  Difference in cost-effectiveness of offering cervical cancer screening between both arms. This includes the cost of screening and follow-up visits in primary care, the cost of further investigations in primary and tertiary care and the cost of treatment for CIN and cervical cancer in tertiary care.
Facilitators and barriers of uptake of cervical cancer screening | 1 year
  Assessing the factors associated with uptake of cervical cancer screening. These factors include demographics of participants (age, ethnicity, education level, marital status, housing type, employment status), Body Mass Index, obstetrics-related factors (menopausal status, pregnancies, previous cervical cancer screening tests, use of tampons or menstrual cups, previous HPV vaccinations) as well as beliefs and attitudes towards cervical cancer screening. These variables will be collected from questionnaires.
Feasibility of self-sampling cervical cancer screening | 1 year
  Assessing the preferences for next screening and the experience of the sampling procedure (ease of conducting, comfort, anxiety, embarrassment, unpleasantness and trusting of results) from questionnaires.
Risk factors for cervical cancer and CIN | 2 years
  Assessing the factors associated with cervical cancer and CIN. These factors include demographics of participants, family history of cervical cancer, smoking status, use of contraceptives, immunosuppressive conditions and sexual history and obstetrics-related factors. These variables will be collected from questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ng Xin Rong, MBBS, Principal Investigator — National Healthcare Group Polyclinics
Locations (1):
- National Healthcare Group Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng XR, Quek IP, Pereira MJ, Molina JA, Ngeow J, Wong SKW. Randomised controlled trial evaluating the impact of different methods of HPV DNA testing for cervical cancer screening in Singapore's primary care settings: a study protocol. BMJ Open. 2025 Mar 24;15(3):e095091. doi: 10.1136/bmjopen-2024-095091. PMID 40132819